CLINICAL TRIAL: NCT01803698
Title: MANAGEMENT OF GESTATIONAL WEIGHT GAIN BY FAMILY PHYSICIANS: SEEKING CONGRUENCE WITH GUIDELINES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: never started
Sponsor: Helena Piccinini (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Helena Piccinini, Family Physician, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P20PiccVall
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Gestational Weight Gain
Keywords: Pregnancy; Gestational weight gain; Primary care; Guidelines
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training in the use of IOM charts (Experimental): Training family physicians to regularly refer to the Institute of Medicine guideline trajectories and provide feedback about GWG ("training in the use of IOM charts") during routine prenatal visits.
  Interventions: Behavioral: Training in the use of IOM charts
- Usual care (No Intervention): Family physicians providing usual prenatal care.

INTERVENTIONS:
Behavioral: Training in the use of IOM charts
  Arms: Training in the use of IOM charts

SUMMARY:
Background The Institute of Medicine (IOM) published guidelines in 2009 for optimal gestational weight gain (GWG) during pregnancy. These guidelines include trajectories for optimal GWG, based on a woman's pre-pregnancy body mass index (BMI), to be used throughout the duration of a pregnancy. Although there is a significant association between the total GWG recommended by these guidelines and maternal and perinatal outcomes, research has demonstrated that only approximately one-third of pregnant women have total GWG within the recommended amounts. Factors known to influence GWG include maternal age, parity, being in a committed relationship and smoking. In addition, recommendations by primary care providers have been shown to influence actual GWG. Women appreciate advice from their primary care providers, however, despite this, there is evidence that many patients report not being advised at all about GWG by their primary care providers.

Relevance Excess weight gain in pregnancy has been shown to be a modifiable risk factor for excess weight in childhood, thus contributing to the intergenerational cycle of obesity. There is an opportunity to interfere with this cycle during the peri-pregnancy period, as women's motivation to engage in behaviour change is elevated and contact with their primary care providers is frequent.

Research Question and Hypothesis What impact does training family physicians to regularly refer to the IOM trajectories and provide feedback about GWG ("training in the use of IOM charts") during routine prenatal visits, compared to usual care, have on congruence of total GWG with IOM guidelines? Null Hypothesis: there is no difference in the congruence of total GWG with IOM guidelines between women whose family physicians were assigned to training in the use of the IOM charts and those whose family physicians were assigned to usual care.

Objectives

The following are the objectives for this study:

1. To compare the congruence of total GWG with IOM guidelines between women whose family physicians were assigned to training in the use of IOM trajectories and those whose family physicians were assigned to usual care.
2. To explore the relationship between other independent variables (maternal age, parity, committed relationship and smoking) and congruence of total GWG with IOM guidelines, for women whose family physicians were assigned to training in the use of IOM trajectories and for those whose family physicians were assigned to usual care.

ELIGIBILITY:
Inclusion Criteria:

* family physicians who provide prenatal care
* pregnant women with low risk pregnancy

Exclusion Criteria:

* pregnant women < 18 years old
* pregnant women with multiple gestation
* pregnant women with chronic disease
* pregnant women initially presenting in second trimester or later.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Congruence with gestational weight gain guidelines | up to 38 weeks after enrolment
  The congruence of total gestational weight gain with Institute of Medicine guidelines based on pre-pregnancy body mass index.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Piccinini-Vallis, MSc MD, Principal Investigator — Department of Family Medicine Dalhousie University
Locations (1):
- Halifax Regional Municipality, Halifax, Nova Scotia, Canada